CLINICAL TRIAL: NCT02934009
Title: Dermal Profile Analysis Using NMR-MOUSE (Nuclear Magnetic Resonance - Mobile Universal Surface Explorer)
Brief Title: Dermal Profile Analysis Using the NMR-MOUSE
Acronym: SHN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Institute for Technical and Macromolecular Chemistry, RWTH Aachen University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-014
Record Dates: First submitted 2016-09-30; First posted 2016-10-14 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Exposure to Magnetic Field; Hypotension During Dialysis; Disturbance; Balance, Fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialysis patients (Experimental): In this group dialysis patients are measured by NMR-Mobile Universal Surface Explorer® (NMR-Mouse) during their routine dialysis sessions. After a 5 min rest period the arm of the patients is placed onto the NMR-Mouse and measured before the beginning of dialysis. The arm examined is not the shunt arm. The area selected should not display any signs of skin disease or scars from previous surgeries. After the dialysis the same area is measured again in a second measurement. The measurement will be repeated on three different days with each patient.
  Interventions: Device: Dermal nuclear magnetic resonance (NMR)-profile measurement
- Healthy volunteers (Experimental): In this group "kidney-healthy" volunteers will be examined by NMR-Mobile Universal Surface Explorer® (NMR-Mouse) at three different days. The right/left arm or leg will be used for repeated measurement. Altogether 2 measurements per day are reformed in order to evaluate the reproducibility and variability.
  Interventions: Device: Dermal nuclear magnetic resonance (NMR)-profile measurement

INTERVENTIONS:
Device: Dermal nuclear magnetic resonance (NMR)-profile measurement — Nuclear magnetic resonance (NMR)-profile measurement of the dermis
  Other Names: NMR-MOUSE

SUMMARY:
The determination of fluid status in dialysis patients is a major clinical problem. In this study the NMR-MOUSE is used to determine if it can be used to non-invasively determine hydration status of the skin. This evaluation will be performed in dialysis patients and healthy volunteers.

DETAILED DESCRIPTION:
Excretion of urine is impaired in terminal chronic kidney disease patients often requiring dialysis. Fluid management of dialysis patients is solely based on body weight differences before and after dialysis. Patients can suffer from either hypotension if too much fluid is eliminated by dialysis or from fluid-overload symptom (e.g. shortness of breath, edema) if not enough fluid is eliminated.

In this study a mobile non-invasive NMR-MOUSE setup (a nuclear magnetic resonance spectroscopy measurement) is used to measure the hydration status of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Dialysis
* ability to perform NMR-measurement
* Eligibility to sign informed consent
* signed informed consent

Exclusion Criteria:

* implanted cardiac device
* implanted cranial device
* implanted cochlea device
* intrauterine device
* other metallic implants
* tattoo, any skin disease or scars from surgery (in the area of measurement)
* previous skin treatment with cosmetics (of any kind) 24 hours prior to measurement
* wearing of earrings, piercings or hearings-aids during measurement
* participation in other clinical trials 30 days prior to participation in the SHN study
* no written informed consent
* any conditions, as determined by the examiner, that excludes the patient from participation in the study
* subjects with legal guardian
* pregnancy or lactation (a possible pregnancy of a participant before menopause will be excluded before inclusion in the study)
* subjects under employment or with any relation to the the sponsor or the investigator
* participation in any other study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the diffusion coefficient D [m²/s] by NMR-MOUSE in dialysis patients and healthy volunteers | 30 minutes
  The skin will be subjected to a weak magnetic field (B0). The transversal relaxation time T2 [in s] will be measured stepwise in mm (millimeter) profiles for up to 16 mm depth in the skin. From the different measurements per profile of the skin a diffusion coefficient D [m²/s] will be calculated, which changes dependent on the hydration status of the skin.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of NMR-Mouse dermal measurement | 30 minutes
  The overall number of participants with treatment-related adverse events during the study will be investigated.
Time needed for NMR-Mouse dermal measurement | 30 minutes
  The overall time needed to measure each participant of the study will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Floege, M.D., Principal Investigator — RWTH Aachen University
Locations (1):
- University Hospital of RWTH Aachen, Department of Medicine II, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perlo J, Casanova F, Blumich B. Profiles with microscopic resolution by single-sided NMR. J Magn Reson. 2005 Sep;176(1):64-70. doi: 10.1016/j.jmr.2005.05.017. PMID 15975840
- [Background] Danieli E, Blumich B. Single-sided magnetic resonance profiling in biological and materials science. J Magn Reson. 2013 Apr;229:142-54. doi: 10.1016/j.jmr.2012.11.023. Epub 2012 Dec 8. PMID 23290626
- [Background] Perlo J, Casanova F, Blumich B. Single-sided sensor for high-resolution NMR spectroscopy. J Magn Reson. 2006 Jun;180(2):274-9. doi: 10.1016/j.jmr.2006.03.004. Epub 2006 Mar 31. PMID 16580238
- [Background] Medrano G, Eitner F, Floege J, Leonhardt S. A novel bioimpedance technique to monitor fluid volume state during hemodialysis treatment. ASAIO J. 2010 May-Jun;56(3):215-20. doi: 10.1097/MAT.0b013e3181d89160. PMID 20404719
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362